CLINICAL TRIAL: NCT07400640
Title: Which Is More Effective in the Treatment of Postherpetic Neuralgia: Erector Spinae Plane Block or Transcutaneous Radiofrequency?
Brief Title: Erector Spinae Plane Block Versus Transcutaneous Radiofrequency in Postherpetic Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Other Study IDs: ESP Block & Transcutaneous PRF
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postherpetic Neuralgia; Neuropathic Pain; Herpes Zoster
Keywords: postherpetic neuralgia, esp block,transcutaneous rf,
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia; Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erector Spinae Plane Block: Patients with postherpetic neuralgia who received ultrasound-guided erector spinae plane block as part of routine clinical care.
  Interventions: Procedure: Erector Spinae Plane Block
- Transcutaneous Radiofrequency: Patients with postherpetic neuralgia who received transcutaneous radiofrequency treatment applied adjacent to the lesion area as part of routine clinical care
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — 1. Ultrasound-guided erector spinae plane block performed under sterile conditions as part of routine clinical care. After skin antisepsis, a 22-G spinal needle was advanced to the erector spinae plane at the level corresponding to the affected dermatome, and a total volume of 10 mL consisting of dexamethasone, bupivacaine, and normal saline was injected. Patients were observed post-procedure according to standard clinical practice.
  2. Transcutaneous radiofrequency treatment applied adjacent to the affected dermatome as part of routine clinical care. Adhesive surface electrodes were placed over the painful area, and pulsed electrical stimulation was delivered by the device for 10 minutes per session. The procedure was performed once weekly for two sessions, without any modification for research purposes.
  Other Names: Transcutaneous Radiofrequency

SUMMARY:
This observational study aims to compare the effectiveness of ultrasound-guided erector spinae plane (ESP) block and transcutaneous radiofrequency (RF) treatment in patients with postherpetic neuralgia. Pain intensity and neuropathic pain characteristics will be evaluated using the Visual Analog Scale (VAS) and the Self-Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) score.

DETAILED DESCRIPTION:
Postherpetic neuralgia is a challenging neuropathic pain condition that significantly affects quality of life. In routine clinical practice, patients are treated with either ultrasound-guided erector spinae plane block or transcutaneous radiofrequency therapy based on clinician preference and experience.

This observational study includes patients who have already completed one of these treatments as part of standard care in the Algology Clinic. No randomization or modification of treatment plans was performed for research purposes. Patients will be divided into two cohorts according to the treatment they received. Treatment outcomes will be retrospectively evaluated and compared using VAS and S-LANSS scores before treatment, immediately after treatment, and at 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of postherpetic neuralgia involving cervical, thoracic, or lumbar regions

Age between 18 and 80 years

Persistent pain despite conservative treatment

Baseline VAS score > 5

Exclusion Criteria:

Ophthalmic or extremity postherpetic neuralgia

Allergy to local anesthetics

Pregnancy

Coagulopathy or use of antiplatelet therapy

Cognitive impairment preventing informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 80 years diagnosed with postherpetic neuralgia involving cervical, thoracic, or lumbar dermatomes who underwent either ultrasound-guided erector spinae plane block or transcutaneous radiofrequency treatment as part of routine clinical care. Patients were included if they had persistent pain despite conservative treatment and a baseline Visual Analog Scale (VAS) score greater than 5. All treatments were completed prior to study enrollment, and no changes were made to clinical management for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
VAS | Baseline, post-procedure 1 month
  Pain intensity assessed by Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
S-LANSS | Baseline, post-procedure 1 month
  Neuropathic pain severity assessed by S-LANSS score

CONTACTS AND LOCATIONS:
Overall Officials: AYSE BETUL ACAR, Principal Investigator — Diskapi TRH
Locations (1):
- Ayse Betul Acar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No